CLINICAL TRIAL: NCT06660667
Title: A Phase 1/2 Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, and Efficacy of One-time Intravitreal Dose of SAR402663 in Participants With Neovascular Age-related Macular Degeneration
Brief Title: A Safety and Efficacy Study of One-time SAR402663 in Adults With Neovascular Age-related Macular Degeneration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFI17940; U1111-1299-1827 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Part I is nonrandomized sequential dose escalation and Part II is randomized parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part I is an open-label study. Part II is partially masked in which participants, Investigators, and outcomes assessors including reading center (RC) are masked to study intervention. The Sponsor is not masked. Masking will be maintained until all participants reach 52 weeks of follow up after SAR402663 dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part I - SAR402663 open-label (OL) (Experimental): Participants will receive a single dose of SAR402663 on Day 1. Multiple dose levels of SAR402663 will be evaluated in successive cohorts of participants.
  Interventions: Biological: SAR402663; Drug: Diluent
- Part II - SAR402663 Dose A (Experimental): Participants will receive a single dose of SAR402663 on Day 1.
  Interventions: Biological: SAR402663; Drug: Diluent
- Part II - SAR402663 Dose B (Experimental): Participants will receive a single dose of SAR402663 on Day 1.
  Interventions: Biological: SAR402663; Drug: Diluent

INTERVENTIONS:
Biological: SAR402663 — Pharmaceutical form:Liquid formulation-Route of administration:Intravitreal injection
Drug: Diluent — Pharmaceutical form:Liquid solution-Route of administration:Intravitreal injection

SUMMARY:
This is a Phase 1/Phase 2 multicenter study to evaluate the safety and efficacy of a one-time single-eye intravitreal dose of SAR402663 in participants with neovascular age-related macular degeneration.

Participants will be enrolled in one of 2 parts:

* In Part I (dose escalation), multiple dose levels of SAR402663 will be evaluated in successive cohorts of participants
* In Part II (dose expansion), participants will be randomized to receive one of two dose levels selected based on data from Part I. Participants, investigators and outcomes assessors will be masked to dose.

After receiving one-time dose of SAR402663, participants will undergo regular assessments over 12 months. Following this, participants will enter an extended follow-up (EFU) phase for the assessment of safety and durability of clinical activity of SAR402663 through Year 5.

ELIGIBILITY:
Inclusion Criteria:

* Between 50 and 90 years of age
* Participants with diagnosis of macular neovascularization secondary to age-related macular degeneration (nAMD)
* Study eye with best corrected visual acuity (BCVA) ETDRS Snellen equivalent for dose escalation (Part I) between 20/32 and 20/400 and for expansion (Part II) between 20/25 and 20/200
* Current or previous use of anti-vascular endothelial growth factor (VEGF) treatment in the study eye
* Demonstrated a response to anti-VEGF treatment

Exclusion Criteria:

* Any condition in the study eye that may prevent visual acuity improvement or interfere with ocular safety or efficacy assessments
* History of active ocular infection in the study eye in 6 months prior to screening
* Active uncontrolled glaucoma in the study eye
* History of uveitis in either eye
* Current use of ocular corticosteroids in the study eye
* Previous gene therapy
* Any significant poorly controlled illness that would preclude study compliance and follow up

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2027-05-18 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular treatment emergent adverse event (TEAEs) | Day 1 to Week 52
Incidence and severity of ocular treatment emergent serious adverse event (TESAEs) | Day 1 to Week 52
Incidence and severity of non-ocular TEAEs | Day 1 to Week 52
Incidence and severity of non-ocular TESAEs | Day 1 to Week 52
Number of participants with any clinically significant changes in laboratory variables | Day 1 to Week 52
Number of participants with any clinically significant changes in vital signs | Day 1 to Week 52

SECONDARY OUTCOMES:
Percentage of participants not requiring supplemental anti-vascular endothelial growth factor (VEGF) therapy | Day 1 to Week 52 and Week 8 to Week 52
Annualized injection rates of anti-VEGF therapy | Day 1 to Week 52
Change from baseline in BCVA using the ETDRS letter score | Baseline, Week 52
  Visual function of the study eye was assessed at a distance of 4 meters using the best corrected visual acuity (BCVA) early treatment diabetic retinopathy study (ETDRS) letter score. BCVA scale range is 0 (worst score) to 100 (best score).
Percentage of participants not losing more than or equal to 15 ETDRS letters from baseline | Baseline, Week 52
Change from baseline in central subfield thickness (CST), measured by spectral domain optical coherence tomography (SD-OCT) | Baseline, Week 52

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Site # 8400011, Phoenix, Arizona
  - Site # 8400028, Scottsdale, Arizona
  - Site # 8400023, Beverly Hills, California
  - Site # 8400004, Gainesville, Florida
  - Site # 8400002, St. Petersburg, Florida
  - Site # 8400010, Augusta, Georgia
  - Site # 8400005, Lemont, Illinois
  - Site # 8400003, Hagerstown, Maryland
  - Site # 8400009, Boston, Massachusetts
  - Site # 8400021, Reno, Nevada
  - Site # 8400017, Eugene, Oregon
  - Site # 8400016, Ladson, South Carolina
  - Site # 8400018, Germantown, Tennessee
  - Site # 8400008, Abilene, Texas
  - Site # 8400015, Austin, Texas
  - Site # 8400007, Austin, Texas
  - Site # 8400006, Dallas, Texas
  - Site # 8400030, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DFI17940 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26380&tenant=MT_SNY_9011